CLINICAL TRIAL: NCT00571155
Title: Prospective Trial of Intravenous Levetiracetam in Patients With Primary Brain Tumors and at Least One Symptomatic Seizure Who Undergo Biopsy or Cytoreductive Surgery (HELLO-study)
Brief Title: Trial of Levetiracetam in Patients With Primary Brain Tumors and Symptomatic Seizures Who Undergo Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Prof. Michael Weller, University Hospital Tuebingen, Department of General Neurology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HELLO-Study 2007; EudraCT Number: 2007-005063-96
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Last update posted 2009-08-20 (Estimated); Status verified 2009-08

CONDITIONS: Primary Brain Tumor; Epilepsy
MeSH Terms: conditions — Brain Neoplasms; Epilepsy | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Drug: levetiracetam

INTERVENTIONS:
Drug: levetiracetam — oral and intravenous dosing 2000-3000 mg per day
  Other Names: Keppra

SUMMARY:
The purpose of this study is to determine the feasibility, efficacy and safety of intravenous and oral antiepileptic treatment with levetiracetam in patients with primary brain tumors and symptomatic epilepsy in the period of neurosurgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* suspected primary brain tumor by imaging
* planned bioptical or cytoreductive surgery of the tumor
* symptomatic epilepsy
* Karnofsky performance score ≥ 70%
* women with child bearing potential must perform sufficient contraception
* sufficient haematologic, hepatic and renal function by laboratory testing

Exclusion Criteria:

* treatment with other antiepileptic drugs other than levetiracetam in the last seven days before surgery
* known allergic reaction to levetiracetam or other serious side effects
* known, not tumor-induced, epilepsy
* previous brain surgery
* dementia
* participation in another clinical trial
* addiction to drugs or alcohol
* pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Feasibility of standardized treatment of patients with primary brain tumors and symptomatic epilepsy with levetiracetam in the period of neurosurgical intervention. | 1 year

SECONDARY OUTCOMES:
Efficacy, safety and tolerance of intravenous and oral levetiracetam in patients with primary brain tumors and symptomatic epilepsy in the period of neurosurgical intervention. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael Weller, MD, Principal Investigator — University-Hospital of Tuebingen, Department of General Neurology
Locations (1):
- University Hospital Tuebingen, Department of General Neurology, Tübingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Derived] Bahr O, Hermisson M, Rona S, Rieger J, Nussbaum S, Kortvelyessy P, Franz K, Tatagiba M, Seifert V, Weller M, Steinbach JP. Intravenous and oral levetiracetam in patients with a suspected primary brain tumor and symptomatic seizures undergoing neurosurgery: the HELLO trial. Acta Neurochir (Wien). 2012 Feb;154(2):229-35; discussion 235. doi: 10.1007/s00701-011-1144-9. Epub 2011 Sep 10. PMID 21909835